CLINICAL TRIAL: NCT06378866
Title: MC230502 Dynamic Investigator Initiated Enterprise (DIVINE) in Prostate Cancer
Brief Title: Stereotactic Body Radiation Therapy Plus Immediate or Delayed Androgen Receptor Pathway Inhibitor and Androgen Deprivation Therapy or Salvage Radiation Therapy for the Treatment of Prostate Cancer, DIVINE Trial
Acronym: DIVINE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC230502; R01CA286127 (NIH); NCI-2024-02978 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23-012176 (Other: Mayo Clinic Institutional Review Board); MC230502 (Other: Mayo Clinic in Rochester)
Record Dates: First submitted 2024-04-16; First posted 2024-04-23 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Recurrent Castration-Sensitive Prostate Carcinoma; Recurrent Prostate Cancer; Castration-resistant Prostate Cancer; Biochemically Recurrent Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — abiraterone; Abiraterone Acetate; apalutamide; Specimen Handling; darolutamide; acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; enzalutamide; Goserelin; histrelin; Leuprolide; Magnetic Resonance Spectroscopy; X-Rays; Watchful Waiting; Observation; Prednisone; deltacortene; prednylidene; relugolix; Radiosurgery; Triptorelin Pamoate; Radiotherapy; Radiation; Radiotherapy, Image-Guided

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group A (SBRT, APRI, ADT) (Active Comparator): Patients undergo SBRT and receive ARPI (abiraterone and prednisone, apalutamide, darolutamide, or enzalutamide) and ADT (leuprolide, triptorelin, histrelin, goserelin, degarelix, or relugolix). Cycles repeat every 4 months (16 weeks) for up to 6 months in the absence of unacceptable toxicity. Patients then undergo watchful waiting thereafter until disease progression. Additionally, patients undergo blood sample collection and PET, CT, MRI, or bone scan throughout the trial.
  Interventions: Drug: Abiraterone; Drug: Apalutamide; Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Drug: Darolutamide; Drug: Degarelix; Drug: Enzalutamide; Drug: Goserelin; Drug: Histrelin; Drug: Leuprolide; Procedure: Magnetic Resonance Imaging; Other: Patient Observation; Procedure: Positron Emission Tomography; Drug: Prednisone; Other: Questionnaire Administration; Drug: Relugolix; Radiation: Stereotactic Body Radiation Therapy; Drug: Triptorelin
- Group B (SBRT, watchful waiting) (Experimental): Patients undergo SBRT with watchful waiting. Cycles repeat every 4 months (16 weeks) in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection and PET, CT, MRI, or bone scan throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Other: Patient Observation; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Radiation: Stereotactic Body Radiation Therapy; Radiation: Radiation Therapy
- Group C (sXRT, watchful waiting) (Experimental): Patients undergo sXRT with watchful waiting. Cycles repeat every 4 months (16 weeks) in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection and PET, CT, MRI, or bone scan throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Other: Patient Observation; Procedure: Positron Emission Tomography; Other: Questionnaire Administration
- Group D (initial observation, image-guided therapy) (Active Comparator): Patients undergo initial observation with subsequent image-guided therapy based on visualized distant progression, which may consist of cross-over to groups A & B, other off-trial radiotherapy, systemic therapy, surgical intervention, or other intervention per clinician discretion. Cycles repeat every 4 months (16 weeks) in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo blood sample collection and PET, CT, MRI, or bone scan throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Other: Patient Observation; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Procedure: Image-Guided Therapy

INTERVENTIONS:
Drug: Abiraterone — Given abiraterone
  Other Names: Abiraterone acetate; CB-7598; CB7598; Zytiga
  Arms: Group A (SBRT, APRI, ADT)
Drug: Apalutamide — Given apalutamide
  Other Names: ARN 509; ARN-509; ARN509; Erleada; JNJ 56021927; JNJ-56021927
  Arms: Group A (SBRT, APRI, ADT)
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Scan — Undergo bone scan
  Other Names: Bone Scintigraphy
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography (CAT); Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Drug: Darolutamide — Given darolutamide
  Other Names: Antiandrogen ODM-201; BAY 1841788; BAY-1841788; BAY1841788; Nubeqa; ODM 201; ODM-201
  Arms: Group A (SBRT, APRI, ADT)
Drug: Degarelix — Given degarelix
  Other Names: ASP3550; FE200486; Firmagon
  Arms: Group A (SBRT, APRI, ADT)
Drug: Enzalutamide — Given enzalutamide
  Other Names: ASP9785; MDV3100; Xtandi
  Arms: Group A (SBRT, APRI, ADT)
Drug: Goserelin — Given goserelin
  Other Names: ICI-118630
  Arms: Group A (SBRT, APRI, ADT)
Drug: Histrelin — Given histrelin
  Arms: Group A (SBRT, APRI, ADT)
Drug: Leuprolide — Given leuprolide
  Other Names: Leuprorelin
  Arms: Group A (SBRT, APRI, ADT)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; Nuclear Magnetic Resonance (NMR) Imaging; NMRI; Nuclear Magnetic Resonance Imaging (NMRI); sMRI; Structural MRI (sMRI); NMR Imaging
Other: Patient Observation — Undergo watchful waiting or initial observation
  Other Names: Active Surveillance; deferred therapy; expectant management; Observation; Watchful Waiting
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography (PET); Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Drug: Prednisone — Given prednisone
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
  Arms: Group A (SBRT, APRI, ADT)
Other: Questionnaire Administration — Ancillary studies
Drug: Relugolix — Given relugolix
  Other Names: N-(4-(1-((2,6-Difluorophenyl)methyl)-5-((dimethylamino)methyl)-1,2,3,4-tetrahydro-3-(6-methoxy-3-pyridazinyl)-2,4-dioxothieno(2,3-d)pyrimidin-6-yl)phenyl)-N'-methoxyurea; Orgovyx; Relumina; TAK 385; TAK-385
  Arms: Group A (SBRT, APRI, ADT)
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation (SABR); Stereotactic Ablative Body Radiation Therapy
  Arms: Group A (SBRT, APRI, ADT); Group B (SBRT, watchful waiting)
Drug: Triptorelin — Given triptorelin
  Other Names: 6-D-Tryptophan-LH-RH; 6-D-Tryptophanluteinizing Hormone-releasing Factor; AY-25650; AY25650; CL-118,532; CL118532; Detryptoreline
  Arms: Group A (SBRT, APRI, ADT)
Radiation: Radiation Therapy — Undergo sXRT
  Other Names: Cancer Radiotherapy; Irradiation; RADIATION; Radiotherapeutics; RADIOTHERAPY
  Arms: Group B (SBRT, watchful waiting)
Procedure: Image-Guided Therapy — Undergo image-guided therapy
  Other Names: Image Guided Therapy
  Arms: Group D (initial observation, image-guided therapy)

SUMMARY:
This phase II trial studies the effects of stereotactic body radiation therapy (SBRT) and the timing of treatment with androgen receptor pathway inhibitor (ARPI) plus androgen deprivation therapy (ADT) in treating patients with hormone sensitive prostate cancer that has spread from where it first started to other places in the body (metastatic), and that has come back after a period of improvement (recurrent). It also studies the effects of salvage radiation therapy (sXRT) on prostate cancer and to see if radiation to the pelvis helps prevent prostate cancer from spreading elsewhere. SBRT is a type of external radiation therapy that uses special equipment to position a patient and precisely deliver radiation to tumors in the body (except the brain). The total dose of radiation is divided into smaller doses given over several days. This type of radiation therapy helps spare normal tissue. Androgen can cause the growth of prostate cells. ADT lowers the amount of androgen made by the body. This may help stop the growth of tumor cells that need androgen to grow. Androgen receptor pathway inhibitors work by blocking the effects of androgen to stop the growth and spread of tumor cells. sXRT is a targeted radiation treatment for the prostate, typically given when cancer possibly returns after surgery or radiation. Its goal is to destroy any tumor cells in the area. Giving SBRT alone with watchful waiting may be as effective in treating prostate cancer as giving SBRT together with ARPI and ADT and sXRT may be effective in treating prostate cancer and preventing it from spreading elsewhere.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate and compare modified radiographic progression-free survival (mrPFS) in patients with metachronous recurrent oligometastatic prostate cancer treated with SBRT and 6 months ADT/ARPI followed by watchful wait (Group A) versus SBRT followed by watchful waiting (Group B). (De-escalation stratified by Extracellular Vesicles--Irradiation with Antiandrogen Therapy Exclusion [DEVIATE]) II. To evaluate and compare distant progression-free survival (PFS), landmarked at 12 months, in patients with biochemically recurrent prostate cancer treated with sXRT followed by watchful waiting (Group C) versus initial observation and subsequent image-guided therapy (Group D). (Biochemical Recurrence Irradiation versus Observation [BRIO])

SECONDARY OBJECTIVES:

I. To evaluate and compare overall survival (OS) between treatment groups. II. To evaluate and compare biochemical progression-free survival (bPFS) between treatment groups.

III. To evaluate and compare distant progression-free survival (PFS) starting from study registration, in patients with biochemically recurrent prostate cancer treated with sXRT followed by watchful waiting (Group C) versus initial observation and subsequent image-guided therapy (Group D).

TERTIARY OBJECTIVES:

I. To estimate rates of salvage radiotherapy to the pelvis in patients with biochemically recurrent prostate cancer treated with initial observation and subsequent image-guided therapy (Group D).

II. To evaluate the adverse event profile of the study treatments as assessed per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE).

III. To evaluate and compare castration-resistant prostate cancer (CRPC)-free survival between treatment groups NOTE: CRPC-free survival: radiographic progression-free survival with castrate-level testosterone (< 50ng/mL).

IV. Determine the efficacy of extracellular vesicles (EVs) as a minimal residual disease (MRD) marker.

V. Determine the efficacy of EVs as an early indicator of disease relapse. VI. Determine whether early ADT and ARPI hasten CRPC. VII. Determine how circulating tumor deoxyribonucleic acid (ctDNA) compares as a biomarker to EVs.

OUTLINE: Patients are assigned to 1 of 2 cohorts.

DEVIATE COHORT: Patients are randomized to 1 of 2 groups.

GROUP A: Patients undergo SBRT and receive ARPI (abiraterone and prednisone, apalutamide, darolutamide, or enzalutamide) and ADT (leuprolide, triptorelin, histrelin, goserelin, degarelix, or relugolix). Cycles repeat every 4 months (16 weeks) for up to 6 months in the absence of disease progression or unacceptable toxicity. Patients then undergo watchful waiting thereafter until disease progression.

GROUP B: Patients undergo SBRT with watchful waiting. Cycles repeat every 4 months (16 weeks) in the absence of disease progression or unacceptable toxicity.

BRIO COHORT: Patients are randomized to 1 of 2 groups.

GROUP C: Patients undergo sXRT with watchful waiting. Cycles repeat every 4 months (16 weeks) in the absence of disease progression or unacceptable toxicity.

GROUP D: Patients undergo initial observation with subsequent image-guided therapy based on visualized distant progression, which may consist of cross-over to groups A & B, other off-trial radiotherapy, systemic therapy, surgical intervention, or other intervention per clinician discretion. Cycles repeat every 4 months (16 weeks) in the absence of disease progression or unacceptable toxicity.

Additionally, all patients undergo blood sample collection and positron emission tomography (PET), computed tomography (CT), magnetic resonance imaging (MRI), or bone scan throughout the trial.

Upon completion of study interventions patients are followed up every 6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Disease characteristics:

  * DEVIATE (Groups A and B only):

    * Clinical confirmation of metachronous (metastatic) recurrent hormone-sensitive prostate cancer
    * Five (5) or fewer metastases with at least one metastasis beyond the pelvis on advanced molecular and/or conventional imaging
    * Serum testosterone > 100ng/dL
  * BRIO (Gropus C & D only):

    * Prostate-specific antigen (PSA) between 0.2 and 1.5 ng/mL with PSA above 0.2 on at least two consecutive measurements at least 5 days apart
    * No local or metastatic recurrence apparent on advanced molecular imaging
    * Serum testosterone > 100 ng/dL
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0, 1 or 2
* Hemoglobin ≥ 8.0 g/dL (obtained ≤ 15 days prior to registration)
* Absolute neutrophil count (ANC) ≥ 1500/mm^3 (obtained ≤ 15 days prior to registration)
* Platelet count ≥ 80,000/mm^3 (obtained ≤ 15 days prior to registration)
* Alanine aminotransferase (ALT) and aspartate transaminase (AST) ≤ 3 x upper limit of normal (ULN) ( ≤ 5 x ULN for patients with liver involvement) (obtained ≤ 15 days prior to registration)
* Calculated creatinine clearance ≥ 30 ml/min using the Cockcroft-Gault formula (obtained ≤ 15 days prior to registration)
* Provide written informed consent
* Ability to complete questionnaire(s) by themselves or with assistance
* Willingness to provide mandatory blood specimens for correlative research
* Willingness to provide tissue specimens for correlative research
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)

Exclusion Criteria:

* Any of the following because this study involves an investigational agent, the genotoxic, mutagenic, and teratogenic effects of which on the developing fetus and newborn are unknown

  * Pregnant persons
  * Nursing persons
  * Persons of childbearing potential or able to father a child who are unwilling to employ adequate contraception
* Prior metastasis-directed therapy
* Any of the following prior therapies:

  * Surgery ≤ 3 weeks prior to registration
  * Chemotherapy for prostate cancer at any time
  * Androgen receptor pathway inhibitor such as abiraterone, apalutamide, darolutamide, or enzalutamide in the last 2 years
* Uncontrolled intercurrent non-cardiac illness including, but not limited to:

  * Ongoing or active infection
  * Psychiatric illness/social situations
  * Dyspnea at rest due to complications of advanced malignancy or other disease that requires continuous oxygen therapy
  * Any other conditions that would limit compliance with study requirements
* Receiving any other investigational agent which would be considered as a treatment for prostate cancer.
* Failure to recover from acute, reversible effects of prior therapy regardless of interval since last treatment EXCEPTION: Grade 1 peripheral (sensory) neuropathy that has been stable for at least 3 months since completion of prior treatment
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Or psychiatric illness/social situations that would limit compliance with study requirements
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Other active malignancy ≤ 3 years prior to registration

  * EXCEPTIONS: Curatively treated non-melanotic skin cancer or papillary thyroid cancer
  * NOTE: If there is a history of prior malignancy, they must not be receiving other specific treatment such as chemotherapy or antihormonal therapy for their cancer
* History of myocardial infarction ≤ 6 months prior to registration, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 532 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2029-05-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Modified radiographic progression-free survival (mrPFS) (Groups A & B) | Up to 5 years
  Modified radiographic progression-free survival (mrPFS) is defined as the time from the date of randomization (enrollment to study) to the date of the first occurrence of the following events: death due to all causes or radiographic progression per Prostate Cancer Working Group 3 Criteria, which is not addressable by stereotactic body radiation therapy (SBRT). Radiographic progression not addressable by SBRT per the treating physician NOTE: Radiographic progression disease that can be addressed by SBRT will not be an mrPFS event. NOTE: Event-free patients will be censored at their last imaging assessment.
Distant progression-free survival (PFS) (Groups C & D) | Up to 5 years
  Defined as the date from the date of randomization + 1 year to the date of the first occurrence of death due to all causes or distant progression. Local progression will NOT be considered a distant progression event. Event-free patients will be censored at their last imaging assessment or prostate-specific antigen evaluation, whichever is later.

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 5 years
  Defined as time from randomization (enrolled to study) to the date of death due to any cause. Will be conducted on modified intent-to-treat (mITT) and per-protocol (PP) populations whenever it is applicable and plausible. Safety-related analyses will be performed on the safety population.
Biochemcial progression-free survival (bPFS) | Up to 5 years
  Defined as the time from randomization (enrollment to study) up to the date of death due to any cause or biochemical progressive disease, whichever occurs first. Will be conducted on mITT and PP populations whenever it is applicable and plausible. Safety-related analyses will be performed on the safety population.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob J. Orme, MD, PhD, Principal Investigator — Mayo Clinic in Rochester
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Phoenix, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials